CLINICAL TRIAL: NCT05081063
Title: Low-Titer O Positive Whole Blood Versus Component Therapy for Emergent Transfusion in Trauma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kaushik Mukherjee, Head of Surgery, Trauma Division, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5210170
Record Dates: First submitted 2021-06-07; First posted 2021-10-18 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhagic Shock; Acute Blood Loss Anemia; Traumatic Brain Injury
MeSH Terms: conditions — Shock, Hemorrhagic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Adult male patients brought to the emergency department as Level A trauma activations who are receiving emergency blood transfusion
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low Titer O+ Whole Blood (Experimental): Low Titer O+ Whole blood provided to Level A trauma patients
  Interventions: Combination Product: Routine labs
- Component Therapy (Active Comparator): Component Therapy of O+ pRBC and FFP dispatched to trauma bay for level A traumas
  Interventions: Combination Product: Routine labs

INTERVENTIONS:
Combination Product: Routine labs — Routine labs will be performed with CBC, BMP, Fox screen, ROTEM viscoelastic test, PT/INR, PTT and venous lactate for standard of care for all patients.

SUMMARY:
Adult male patients brought to the emergency department as Level A trauma activations who are receiving emergency blood transfusion.

Objectives

1. Evaluate PRBC equivalents transfused in each group in the first 24 hours (Primary outcome)
2. Evaluate total transfusion in each group in the first 24 hours (Secondary Outcome) including breakdown by FFP equivalents, platelet units, and cryoprecipitate
3. Evaluate 6 hour, 24 hour, and hospital mortality (Secondary Outcome)
4. Evaluate ICU outcomes in each group

DETAILED DESCRIPTION:
Based on the results from Cotton et al, median transfusion in the component therapy group was 6 PRBC in the first 24 hours and 4 PRBC equivalents in the whole blood group. The standard deviation (estimated from the interquartile range) was approximately 4. Thus with an expectation of alpha = 0.05 and expected power of 90% to detect a similar 2 unit difference in transfusion volume, a sample size of 190 should be sufficient; thus projected sample size of 200 should be more than adequate. Age range will be 18 years and older, and only males will be included in the study. Expected racial/ethnic distribution will be approximately 60% white, 15% black, 8% Asian, and 18% other race. No actual recruitment will be performed; rather all qualifying patients will be included. Consent waiver is being requested.

b. Objectives

1. Evaluate PRBC equivalents transfused in each group in the first 24 hours (Primary outcome)
2. Evaluate total transfusion in each group in the first 24 hours (Secondary Outcome) including breakdown by FFP equivalents, platelet units, and cryoprecipitate
3. Evaluate 6 hour, 24 hour, and hospital mortality (Secondary Outcome)
4. Evaluate ICU outcomes in each group:

1. ICU length of stay 2. Ventilator days 3. SOFA score on day of ICU discharge 4. Presence of ARDS 5. Presence of TRALI 6. Presence of DVT/PE 7. Necessity for Dialysis 8. Necessity for Tracheostomy 9. Evaluate viscoelastic testing parameters in both groups when sent on arrival in ICU

1. Percentage of patients with EXTEM clotting time > 80 sec 2. Percentage of patients with EXTEM amplitude at 10 min < 40mm and FIBTEM amplitude at 10 min ≤ 10mm 3. Percentage of patients with EXTEM amplitude at 10 min < 40mm and FIBTEM amplitude at 10 min > 10mm 4. Percentage of patients with maximum thrombolysis > 15% 5. Interval analyses to be performed after 6 and 12 months with provision to continue the study out to 24 months.

1. Stopping rule: A statistically significant difference in hospital mortality at 6 months or 12 months

1. If in favor of LTOWB, consideration of trial termination and making LTOWB the primary standard of care for all trauma patients receiving emergency transfusion except for child-bearing age females (unless Rh immunoglobulin can be administered)
2. If in favor of component therapy, consideration of trial termination and making component therapy the primary standard care for all trauma patients receiving emergency transfusion

ELIGIBILITY:
Inclusion Criteria:

* all adult male patients brought into the emergency department as LEVEL A trauma activations who are receiving emergency blood transfusions

Exclusion Criteria:

* Female patients (specifically excluded due to risk of alloimmunization of Rh-negative female patients of childbearing age against Rh-positive blood)
* children
* prisoners
* all patients classified as dead upon arrival to the trauma bay

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams J, Merutka N, Meyer D, Bai Y, Prater S, Cabrera R, Holcomb JB, Wade CE, Love JD, Cotton BA. Safety profile and impact of low-titer group O whole blood for emergency use in trauma. J Trauma Acute Care Surg. 2020 Jan;88(1):87-93. doi: 10.1097/TA.0000000000002498. PMID 31464874
- [Background] Murphy C, Silva de Leonardi N. The use of low-titer group O whole blood is independently associated with improved survival compared to component therapy in adults with severe traumatic hemorrhage. Transfusion. 2021 Apr;61(4):1341-1342. doi: 10.1111/trf.16266. No abstract available. PMID 33831229
- [Background] Seheult JN, Anto V, Alarcon LH, Sperry JL, Triulzi DJ, Yazer MH. Clinical outcomes among low-titer group O whole blood recipients compared to recipients of conventional components in civilian trauma resuscitation. Transfusion. 2018 Aug;58(8):1838-1845. doi: 10.1111/trf.14779. Epub 2018 Aug 30. PMID 30160310
- [Background] Hanna K, Bible L, Chehab M, Asmar S, Douglas M, Ditillo M, Castanon L, Tang A, Joseph B. Nationwide analysis of whole blood hemostatic resuscitation in civilian trauma. J Trauma Acute Care Surg. 2020 Aug;89(2):329-335. doi: 10.1097/TA.0000000000002753. PMID 32744830
- [Background] Cotton BA, Podbielski J, Camp E, Welch T, del Junco D, Bai Y, Hobbs R, Scroggins J, Hartwell B, Kozar RA, Wade CE, Holcomb JB; Early Whole Blood Investigators. A randomized controlled pilot trial of modified whole blood versus component therapy in severely injured patients requiring large volume transfusions. Ann Surg. 2013 Oct;258(4):527-32; discussion 532-3. doi: 10.1097/SLA.0b013e3182a4ffa0. PMID 23979267
- [Derived] Strada AM, Suarez G, Luo-Owen X, Tabrizi MB, Rosenthal MG, Stevens WT, Lum SS, Mukherjee K. Pragmatic O-Positive Whole-blood RandoMizaTion in male trauma Patients (POWeR-MTP). Eur J Trauma Emerg Surg. 2025 Apr 16;51(1):175. doi: 10.1007/s00068-025-02848-0. PMID 40237834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male highest-tier trauma activations randomized in 24 hour blocks
Period: Overall Study
Arm/Group | Low Titer O+ Whole Blood | Component Therapy
Started (Beginning of study) | 52 | 147
Completed | 52 | 147
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This population was all male given the safety constraints listed in the protocol. Baseline data was only collected for patients that survived 24 hours as this was the analyzed group as specified in the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Titer O+ Whole Blood | Component Therapy | Total
Number analyzed (Participants) | 52 | 147 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (13.6) | 42.1 (16.9) | 41.5 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Only male patients included as per safety criteria in protocol
  Participants
    Female | 0 | 0 | 0
    Male | 52 | 147 | 199
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Injury severity score [Mean (Standard Deviation); unit: units on a scale] — Standardized description of injury severity used for trauma patients. Score ranges from 1 to 75 and is comprised of the squares of the the three highest individual anatomic injury scores (AIS) for each injured body area (Head, Face, Spine, Chest, Abdomen/Pelvis, Extremities). Each individual AIS score ranges from 1 to 5, with some body areas (Head, Chest, Abdomen/Pelvis) having a potential score of 6 to indicate an unsurvivable injury. 15 and above is considered severely injured.
  units on a scale | 19.6 (11.7) | 19.3 (12.2) | 19.4 (12.0)
Glasgow Coma Scale in ED [Median (Inter-Quartile Range); unit: units on a scale] — Glasgow Coma Scale is a scale to grade neurologic injury. Range 3-15 with E, V, M subscores. E is eye opening with scores: 4 opening spontaneously, 3 opening to voice, 2 opening to painful stimulus, 1 not opening. V is verbal. 5 normal speech, 4 confused speech, 3 incoherent words, 2 incomprehensible sounds, 1 no speech. M is motor with scores of 6 for following commands, 5 for localizing, 4 for withdrawing, 3 for flexor posturing, 2 for extensor posturing, and 1 for no movement. The score is comprised of the E + V + M scores together.
  units on a scale | 13.5 [3 to 15] | 14.0 [3 to 15] | 14 [3 to 15]
First systolic blood pressure in ED [Mean (Standard Deviation); unit: mm Hg] | 91.2 (50.4) | 98.4 (44.6) | 96.5 (46.2)

OUTCOME MEASURES:

1. Primary Outcome: Packed Red Blood Cells Equivalents Units Transfused (1 Whole Blood Unit Treated as 1 Packed Red Blood Cell Unit and 1 Fresh Frozen Plasma Unit)
Description: assessment of pRBC equivalents transfused in each arm, an increase in HGB by 1g/dl per unit transfused will be considered successful
  A blood draw of 5ml will be obtained and tested to assess HGB level. An increase in HGB by 1g/dl per unit transfused will be considered a successful result.
Time Frame: The total transfusion requirement of packed red blood cells was analyzed for the duration of the inpatient hospitalization for patients surviving at least 24 hours. This time is defined as a time period up to 30 days.
Population: Population of patients surviving 24 hours analyzed for transfusion measures
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Low Titer O+ Whole Blood | Component Therapy
Number analyzed (Participants) | 40 | 123
units | 3.8 (5.6) | 5.7 (6.2)

2. Secondary Outcome: Mortality
Description: Assessment of mortality
  This is a composite measurement which includes the following in order to be assessed as pulseless with no respiratory drive or brain death:
  1. there is no evidence of arousal or awareness to maximal external stimuli
  2. pupils are fixed in a midsized or dilated position and non reactive to light
  3. corneal, oculocephalic and oculovestibular reflexes are absent
  4. There is no facial movement to noxious stimuli
  5. the gag reflex is absent to bilateral posterior pharyngeal stimuli
  6. the cough reflex is absent to deep tracheal suctioning
  7. there is no brain mediated motor response to noxious stimuli of the limbs
  8. spontaneous respirations are not observed when apnea test targets reach pH <7.30 and PaCO2 >60mmhg
Time Frame: In patients surviving at least 24 hours who were included in analysis of outcome measures, we assessed survival to hospital discharge. This means the duration of time in the hospital up to discharge with a maximum of 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Titer O+ Whole Blood | Component Therapy
Number analyzed (Participants) | 40 | 123
Participants | 4 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through hospital discharge, meaning the duration of time in the hospital after the injury up to 30 days.
Arm/Group | Low Titer O+ Whole Blood | Component Therapy
All-Cause Mortality (participants affected / at risk) | 17/52 | 37/147
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/147
Other Adverse Events (participants affected / at risk) | 0/52 | 0/147

LIMITATIONS AND CAVEATS:
Sample size Difference between size of groups Pragmatic randomization scheme

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT05081063/Prot_SAP_001.pdf
  • Study Protocol: Clarification of Study Protocol Date (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05081063/Prot_002.pdf